CLINICAL TRIAL: NCT02943642
Title: Safety and Effectiveness of A-dmDT390-bisFv(UCHT1) Fusion Protein (Resimmune®) in Subjects With Mycosis Fungoides: A Phase II Multi-center Randomized Clinical Trial
Brief Title: Safety and Effectiveness of A-dmDT390-bisFv(UCHT1) Fusion Protein in Subjects With Mycosis Fungoides
Acronym: Resimmune®
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angimmune LLC (Industry)
Collaborators: City of Hope National Medical Center (Other); Columbia University (Other); Dana-Farber Cancer Institute (Other); Northwestern University Feinberg School of Medicine (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Ohio State University Comprehensive Cancer Center (Other); Rush University Medical Center (Other); Scott and White Hospital & Clinic (Other); Yale University (Other); Stanford University (Other); Thomas Jefferson University (Other); University of Arkansas (Other); University of Colorado, Denver (Other); University of Texas Southwestern Medical Center (Other); University of Washington (Other); Vanderbilt University School of Medicine (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FDA IND 100712 Phase II
Record Dates: First submitted 2016-10-18; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Mycosis Fungoides
Keywords: MF; CTCL; Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — A-dmDT390-bisFv(UCHT1) protein; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A-dmDT390-bisFv(UCHT1) (Experimental): A-dmDT390-bisFv(UCHT1) will be administered as Total Dose µg/kg given as 1/8 Total Dose µg/kg/injection twice a day 4-6 hours apart for four consecutive days (days 1-4) into a free flowing IV over a period of approximately 15 minutes.
  Interventions: Biological: A-dmDT390-bisFv(UCHT1)
- Vorinostat (Active Comparator): Subjects in the control arm will receive oral vorinostat capsules at a dose of 400 mg daily up to 12 months in duration until disease progression or uncontrolled side effects take place. Subjects in the vorinostat arm who experience progressive disease may cross over into the experimental arm after 6 months of treatment after a 2-week vorinostat washout period.
  Interventions: Drug: Vorinostat
- Lead-in Dosing single arm (Experimental): Dose Group 1: A-dmDT390-bisFv(UCHT1) will be administered as 5 µg/kg given as 0.625 µg/kg/injection twice a day 4-6 hours apart for four consecutive days (days 1-4) into a free flowing IV over a period of approximately 15 minutes.
  Dose Group 2: A-dmDT390-bisFv(UCHT1) will be administered as 10 µg/kg given as 1.25 µg/kg/injection twice a day 4-6 hours apart for four consecutive days (days 1-4) into a free flowing IV over a period of approximately 15 minutes.
  Interventions: Biological: A-dmDT390-bisFv(UCHT1)

INTERVENTIONS:
Biological: A-dmDT390-bisFv(UCHT1) — anti-T cell immunotoxin (antibody targeting CD3 on T-cells tagged with diphtheria toxin without binding domain)
  Other Names: Resimmune® (proposed marketing designation)
  Arms: A-dmDT390-bisFv(UCHT1); Lead-in Dosing single arm
Drug: Vorinostat — ZOLINZA is a histone deacetylase (HDAC) inhibitor indicated for the treatment of cutaneous manifestations in patients with cutaneous T-cell lymphoma (CTCL) who have progressive, persistent or recurrent disease on or following two systemic therapies.
  Other Names: Zolinza
  Arms: Vorinostat

SUMMARY:
This study evaluates the effectiveness - as judged by complete response - of a single four-day treatment with the fusion protein A-dmDT390-bisFv(UCHT1) compared to oral Zolinza (Vorinostat), in a randomized 2-arm trial after a maximum of 12 months of treatment. Patient eligibility is stage IB/IIB mycosis fungoides with mSWAT < 50 who have never had lymphoid disease or a prior bone marrow / HSCT transplant.

DETAILED DESCRIPTION:
Primary Objective: This study objective is to document the incidence of complete responses compared to oral vorinostat, in a randomized 2-arm trial after a maximum of 12 months of treatment for subjects with stage IB/IIB mycosis fungoides with mSWAT < 50 who have never had lymphoid disease or a prior bone marrow / HSCT transplant.

Secondary Objective: To further explore the toxicity profile of A-dmDT390-bisFv(UCHT1) fusion protein for subjects with mycosis fungoides who have been selected to be free from preexisting cardiac disease and never treated with Campath.

Number of Subjects: Lead-in Dosing: 12 / Randomized: 162

Patients will receive full supportive care during the course of the study. Participation in the study will require IV infusions of the research agent 2 times a day for four days (protocol FDA outpatient approved), as well as frequent outpatient blood draws for the first 30 days. Patients with partial or complete remissions at their 1 month follow up visit will have another follow-up visit on day 60, then every three months for 1 year, followed by annual visits to assess duration of the response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed the current IRB approved informed consent prior to registration (see Informed Consent).
* Mycosis fungoides, confirmed by biopsy or flow cytometry, without large cell transformation.
* Relapse or progression after 2 or more systemic therapies. Note: Total electron beam therapy can be counted as a systemic therapy.
* Disease stage as follows:

  * Stage IB with no lymph node involvement including lymphadenopathy with mSWAT <50;
  * Stage IIB with no lymph node involvement including lymphadenopathy with mSWAT <50.
* Age 18 years.
* Subjects must have a performance status of < 2 on Eastern Cooperative Oncology Group scale (see Appendix A).
* Subjects must have normal lung function evaluated by pulse oximetry with O2 saturation values between 95-100%.
* Subjects must have fully recovered from toxicity of prior chemotherapy or radiation therapy.
* Subjects must have:

  * bilirubin < 1.5 mg/dL,
  * transaminases < 2.5 X ULN,
  * albumin > 3 gm/dL,
  * creatinine < 2.0 mg/dL.
  * Subjects who have had albumin < 3 gm/dL boosted by an albumin infusion must be observed to maintain albumin at > 3gm dL for 14 days without an additional infusion.
* Subjects must have a normal echocardiogram (EF > 50% normal) without any evidence of cardiac chamber hypertrophy, dilatation or hypokinesis.
* Females and males must be willing to use an approved form of birth control while on this study and for 2 weeks after completion.
* Subjects must have a pretreatment anti-DT titer of 20 μg/ml or less. Subjects with titers between 21 and 35 μg/ml will have an additional anti-DT neutralization test using subject's serum and A-dmDT390-bisFv(UCHT1). If neutralization is not found these titers will be considered acceptable.

Exclusion Criteria:

* Failure to meet any of the criteria.
* Inability to give informed consent because of psychiatric problems, or complicated medical problems.
* Allergic to diphtheria toxin a component of the study drug A-dmDT390-bisFv(UCHT1).
* Serious concurrent medical problems, uncontrolled infections, or disseminated intravascular coagulopathy (DIC), hepatic cirrhosis, or chronic kidney disease.
* CNS leukemia.
* Preexisting cardiovascular disease. The only exception being well controlled essential hypertension with a sitting blood pressure (B.P.) of <160 systolic and <90 diastolic without any evidence of structural heart disease or one episode of myocardial infarction > 8 months ago. Subjects receiving a beta-blocker for hypertension should be converted to another antihypertensive drug class 2-3 weeks before receiving the study drug to prevent a drug-drug interaction reactive tachycardia. Angiotensin inhibitors, angiotensin receptor blockers and calcium channel blockers are all acceptable. A past history of any of the following conditions is considered as exclusions to study participation:

  * Congestive heart failure,
  * Atrial fibrillation,
  * Pulmonary hypertension,
  * Anticoagulant drug therapy,
  * Thromboembolic events,
  * Cardiomyopathy or a myocardial infarction within the past 8 months. The PI and the Clinical Coordinator will be asked to verify that their referred subjects do not have these exclusionary histories listed in 3.2 and a copy of this verification must be sent to the Sponsor before the Sponsor will approve of enrollment. Referring physicians will not need to sign.
* Pregnant or nursing women will be excluded from study.
* History of cirrhosis of the liver based on the Child-Pugh score of Class B or C are not eligible to participate.
* Prior treatment with alemtuzumab (Campath) or similar agents or procedures that depress blood T cell counts to below 50% of the lower limit of normal.
* Prior history of bone marrow transplant or HSCT is an exclusion.
* Prior treatment with vorinostat (Prior treatment with vorinostat for lead-in dosing arm is acceptable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Complete Responses (CR) | Skin lesions will be judged for mSWAT scores for judging the duration of response at 12 months in the experimental arm and 6 months in the comparator arm.
  Evaluation of Target Lesions
  Complete Response (CR) in mycosis fungoides: (a) Cutaneous lesions consisting of erythematous patches and plaques and erythroderma must be absent giving an mSWAT of 0 that persists for at least 30 days, and (b) the spleen and liver should be normal sized by physical exam. Subjects in the experimental arm who have a CR at 12 months will be encouraged to enter the Part B followup that consists of a a yearly physical exam from year 2 to year to year 6 and skin assessment as long as the CR is maintained.
  Partial Response (PR) in mycosis fungoides: (a) There must be a reduction of 50% in cutaneous lesions as judged by mSWAT and (b) no new evidence of disease or disease progression of skin lesions.
  Progressive Disease (PD): At least a 25% increase in the mSWAT score from its nadir value.
  Treatment Failure: Failure to achieve a PR or CR: Relapse/Progression: Relapse is defined at reevaluation as no longer a CR or PR.

SECONDARY OUTCOMES:
Progression Free Survival | 12 months
  Determine the Progression Free Survival duration, PFS
Median duration of Complete Response | 12 months
  Determine the Median duration of CR for each arm.

OTHER OUTCOMES:
Primary Toxicity profile | 3 months
  Determine the Primary Toxicity profile for treatment of A-dmDT390-bisFv(UCHT1). Toxicities from the previous phase I clinical trial known to be associated with A-dmDT390-bisFv(UCHT1) include:
  * Frequent: elevated AST, ALT and CPK; hypersensitivity reactions such as rigors and chills during infusions, hypoalbuminemia.
  * Rare: Vascular leak syndrome.
  * Hypersensitivity infusion reaction.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Frankel AE, Woo JH, Ahn C, Foss FM, Duvic M, Neville PH, Neville DM. Resimmune, an anti-CD3epsilon recombinant immunotoxin, induces durable remissions in patients with cutaneous T-cell lymphoma. Haematologica. 2015 Jun;100(6):794-800. doi: 10.3324/haematol.2015.123711. Epub 2015 Mar 20. PMID 25795722
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956